CLINICAL TRIAL: NCT02383043
Title: Impact of Sustained Release d-Amphetamine on Choice Between Cocaine and a Non-Drug Reinforcer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Joshua A. Lile, Ph.D. (Other)
Responsible Party: Sponsor-Investigator, Joshua A. Lile, Ph.D., Joshua A. Lile, Ph.D., Associate Professor of Behavioral Science, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: R01DA033364-02 (NIH)
Record Dates: First submitted 2015-02-27; First posted 2015-03-09 (Estimated); Results first posted 2019-04-11 (Actual); Last update posted 2019-04-11 (Actual); Status verified 2019-03

CONDITIONS: Active Cocaine Users
MeSH Terms: interventions — Cocaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Treatment (Experimental): Cocaine choice during d-amphetamine maintenance
  Interventions: Drug: Cocaine; Drug: Sustained Release d-Amphetamine
- Placebo Treatment (Placebo Comparator): Cocaine choice during placebo maintenance
  Interventions: Drug: Cocaine; Drug: Sustained Release d-Amphetamine

INTERVENTIONS:
Drug: Cocaine
Drug: Sustained Release d-Amphetamine
  Other Names: Dexedrine Spansule SR

SUMMARY:
Cocaine-use disorders continue to be a significant public health concern, yet no effective medications have been identified. The goal of this study is to establish a research platform for the development of medications for treatment of cocaine abuse and dependence. This study will incorporate choice self-administration procedures between drug and a non-drug alternative reinforcer presented during maintenance on d-amphetamine, which has been previously shown to reduce cocaine use.

ELIGIBILITY:
Inclusion Criteria:

* Recent cocaine use, otherwise healthy

Exclusion Criteria:

* Laboratory results outside of clinically acceptable ranges, history of or current serious physical or psychiatric disease

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2018-04-05 (Actual); Study Completion 2018-04-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratory of Human Behavioral Pharmacology, Lexington, Kentucky, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo, 30 mg d-Amphetamine, 60 mg d-Amphetamine: Cocaine choice during placebo, 30 mg d-Amphetamine, 60 mg d-Amphetamine maintenance
  Placebo and Cocaine
  Placebo and Sustained Release d-Amphetamine
- 30 mg d-Amphetamine, Placebo, 60 mg d-Amphetamine: Cocaine choice during 30 mg d-Amphetamine, Placebo, 60 mg d-Amphetamine maintenance
  Placebo and Cocaine
  Placebo Sustained Release d-Amphetamine maintenance
- 30 mg d-Amphetamine, 60 mg d-Amphetamine, Placebo: Cocaine choice during 30 mg d-Amphetamine, 60 mg d-Amphetamine, Placebo maintenance
  Placebo and Cocaine
  Placebo and Sustained Release d-Amphetamine
Period: Overall Study
Arm/Group | Placebo, 30 mg d-Amphetamine, 60 mg d-Amphetamine | 30 mg d-Amphetamine, Placebo, 60 mg d-Amphetamine | 30 mg d-Amphetamine, 60 mg d-Amphetamine, Placebo
Started | 9 | 5 | 4
Completed | 7 | 5 | 4
Not Completed | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 30 mg d-Amphetamine, Placebo, 60 mg d-Amphetamine: Cocaine choice during 30 mg d-Amphetamine, Placebo, 60 mg d-Amphetamine maintenance
  Placebo and Cocaine
  Placebo and Sustained Release d-Amphetamine
- Total: Total of all reporting groups
Arm/Group | Placebo, 30 mg d-Amphetamine, 60 mg d-Amphetamine | 30 mg d-Amphetamine, Placebo, 60 mg d-Amphetamine | 30 mg d-Amphetamine, 60 mg d-Amphetamine, Placebo | Total
Number analyzed (Participants) | 7 | 5 | 4 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 5 | 4 | 16
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 2 | 5
  Male | 5 | 4 | 2 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic/Latino Black Female | 1 | 1 | 0 | 2
  Non-Hispanic/Latino White Female | 1 | 0 | 2 | 3
  Non-Hispanic/Latino Black Male | 3 | 3 | 1 | 7
  Non-Hispanic/Latino White Male | 1 | 1 | 1 | 3
  Hispanic/Latino Black Male | 1 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 5 | 4 | 16

OUTCOME MEASURES:

1. Primary Outcome: The Number of Times Cocaine Was Selected in the Presence of a Monetary Reward Alternative
Description: The reinforcing effects of cocaine were determined using a modified progressive ratio procedure (Lile et al., 2016) in which subjects made 9 choices between each available cocaine dose and money (US$6.00). Reinforcing effects are measured for each cocaine dose during both d-amphetamine and placebo maintenance.
Time Frame: 9 choice trials per cocaine dose level with each trial separated by 30 minutes
Measure: Mean (Standard Error); unit: cocaine choices
Groups:
- 30 mg d-Amphetamine: Cocaine choice during 30 mg d-amphetamine maintenance
  Placebo and Cocaine
  Sustained Release d-Amphetamine
- Placebo Treatment: Cocaine choice during placebo maintenance
  Placebo and Cocaine
  Placebo
- 60 mg d-Amphetamine: Cocaine choice during 60 mg d-amphetamine maintenance
  Placebo and Cocaine
  Sustained Release d-Amphetamine
Arm/Group | 30 mg d-Amphetamine | Placebo Treatment | 60 mg d-Amphetamine
Number analyzed (Participants) | 16 | 16 | 16
cocaine choices
  Placebo Cocaine | 0.06 (0.06) | 0.94 (0.35) | 0.75 (0.36)
  3 mg/70 kg Cocaine | 0.88 (0.43) | 2.50 (0.89) | 0.56 (0.26)
  10 mg/70 kg Cocaine | 1.88 (0.50) | 5.13 (0.93) | 1.50 (0.51)
  30 mg/70kg Cocaine | 4.69 (0.89) | 6.00 (0.99) | 5.19 (0.95)

ADVERSE EVENTS:
Time Frame: 33 days per subject.
Description: Adverse event reporting consists of each the duration of each d-amphetamine maintenance condition as well as during the conduct of a medical safety session in which cocaine doses are administered prior to initiation of d-amphetamine maintenance.
Groups:
- Medical Safety Session: Experimenter administered Placebo and Cocaine delivery. d-Amphetamine maintenance not yet initiated.
- Placebo: Cocaine choice during placebo d-Amphetamine maintenance
  Placebo and Cocaine
- 30 mg d-Amphetamine: Cocaine choice during 30 mg d-Amphetamine maintenance
  Placebo and Cocaine
- 60 mg d-Amphetamine: Cocaine choice during 60 mg d-Amphetamine maintenance
  Placebo and Cocaine
Arm/Group | Medical Safety Session | Placebo | 30 mg d-Amphetamine | 60 mg d-Amphetamine
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18 | 0/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 1/18 | 0/18 | 0/17 | 1/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Medical Safety Session (N=18) | Placebo (N=18) | 30 mg d-Amphetamine (N=17) | 60 mg d-Amphetamine (N=17)
Chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Chest pain after a session with placebo cocaine maintenance on 60 mg d-amphetamine. Cardiovascular monitoring revealed normal vital signs and heart rhythmicity. Pain determined to be musculoskeletal.
Nausea and vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Nausea and vomiting after smoking a cigarette following administration of cocaine doses during the medical safety session.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2017-12-17): https://cdn.clinicaltrials.gov/large-docs/43/NCT02383043/Prot_000.pdf